CLINICAL TRIAL: NCT00316004
Title: Phase 3 Study of Hypertonic Resuscitation Following Severe Traumatic Brain Injury (TBI)
Brief Title: Hypertonic Resuscitation Following Severe Traumatic Brain Injury (TBI)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); U.S. Army Medical Research and Development Command (U.S. Federal Agency); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Department of National Defence (Other Government); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Gerald Van Belle, PhD/Principal Investigator, Resuscitation Outcomes Consortium Data Coordinating Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28226-A - IND 12505; 5U01HL077863-05 (NIH); IND #12505 TBI cohort (Other: FDA)
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Brain Injuries, Traumatic
Keywords: Traumatic; Brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Saline Solution, Hypertonic; Dextrans; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 7.5% hypertonic saline/6% dextran (HSD) (Experimental): 250 ml intravenous bolus administration of 7.5% saline/6% dextran 70
  Interventions: Drug: 7.5% Hypertonic Saline in 6% Dextran-70 (HSD)
- 7.5% hypertonic saline (HS) (Experimental): 250 ml intravenous bolus administration of 7.5% hypertonic saline
  Interventions: Drug: 7.5% Hypertonic Saline (HS)
- 0.9% normal saline (NS) (Placebo Comparator): 250 ml intravenous bolus administration of 0.9% saline
  Interventions: Drug: 0.9% Normal Saline (NS)

INTERVENTIONS:
Drug: 7.5% Hypertonic Saline in 6% Dextran-70 (HSD) — 250 ml intravenous bolus administration of 7.5% saline/6% dextran 70 administered as a one-time bolus fluid for initial resuscitation to injured patients with suspected severe traumatic brain injury in the out-of-hospital setting.
  Other Names: RescueFlo
  Arms: 7.5% hypertonic saline/6% dextran (HSD)
Drug: 7.5% Hypertonic Saline (HS) — 250 ml intravenous bolus administration of 7.5% hypertonic saline administered as a one-time bolus fluid for initial resuscitation to injured patients with suspected severe traumatic brain injury in the out-of-hospital setting.
  Arms: 7.5% hypertonic saline (HS)
Drug: 0.9% Normal Saline (NS) — 250 ml intravenous bolus administration of 0.9% saline administered as a one-time bolus fluid for initial resuscitation to injured patients with suspected severe traumatic brain injury in the out-of-hospital setting.
  Arms: 0.9% normal saline (NS)

SUMMARY:
The purpose of this study is to determine if hypertonic saline with and without dextran can improve neurologic outcomes in victims of severe traumatic brain injury (TBI).

Injury and lost blood from trauma can cause your body to go into shock (low blood pressure related to blood loss). This decreased blood flow can lead to organ damage. In order to restore the blood pressure and blood flow, the medics give fluids into the patients' veins as soon as possible. This is called "resuscitation". The fluid most commonly used is "isotonic" or one that is the same salt concentration as the blood. The investigators are trying to determine if infusing a "hypertonic" fluid or one more concentrated than the blood can increase the blood pressure and restore blood flow more efficiently. The hypertonic fluids they are using are called hypertonic saline with dextran (HSD) and hypertonic saline (no dextran). Hypertonic saline is a salt solution that is slightly more concentrated than blood. Dextran is a sugar solution.

DETAILED DESCRIPTION:
To determine if prehospital administration of 7.5% Hypertonic Saline in 6% Dextran-70 (HSD) OR 7.5% Hypertonic Saline (HS) compared to current standard therapy with NS as an initial resuscitation fluid affects neurological outcome following severe traumatic brain injury.

Trauma is the leading cause of death among North Americans between the ages of 1 and 44 years. The majority of these deaths result from hypovolemic shock or severe brain injury. Patients in hypovolemic shock develop a state of systemic tissue ischemia then a subsequent reperfusion injury at the time of fluid resuscitation. Conventional resuscitation involves the IV administration of a large volume of isotonic or slightly hypotonic (lactated ringers, LR) solutions beginning in the pre-hospital setting. Although not conclusive, prior studies have suggested that alternative resuscitation with hypertonic saline (7.5%) solutions may reduce morbidity or mortality in these patients. Furthermore, hypertonic fluids may have specific advantages in the brain-injured patient, as they may aid in the rapid restoration of cerebral perfusion and prevent extravascular fluid sequestration, thereby limiting secondary brain injury. In addition, recent studies have demonstrated that hypertonicity significantly alters the activation of inflammatory cells, an effect that may reduce subsequent organ injury from ischemia-reperfusion and decrease nosocomial infection.

This study is a randomized, double-blind, three-arm placebo controlled trial designed to evaluate the clinical outcome of trauma patients with severe TBI as manifested by a pre-hospital GCS of 8 or less. Patients will be randomized to a single 250cc IV dose of 7.5% saline in 6% Dextran-70 (HSD), 7.5% saline (HS) or normal saline as the initial fluid for pre-hospital resuscitation. No additional interventions will occur once the patient is admitted to the hospital. In hospital data collection will last up to 28 days. Patients will have neurologic outcome measurements at discharge, 1 month post discharge, and 6 months post injury. Enrollment will be restricted to age ≥ 15 years or ≥ 50 kg if age is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Blunt trauma
* Pre-hospital Glasgow Coma Scale equal to or less than 8(GCS≤8)*
* Age 15 years or older or 50 kg or more

  * Patients who met the inclusion criteria above and did not meet the exclusion criteria below but who had systolic blood pressure (SBP) ≤70 or SBP>70 and SBP≤90 and heart rate (HR)≥108 were included in the Hypertonic Resuscitation following Traumatic Injury study that focused on shock patients who may or may not have a traumatic brain injury (TBI). In other words, patients with both TBI and shock would not be included in this study of TBI patients without shock at the time of enrollment.

Exclusion Criteria:

* Known or suspected pregnancy
* Age younger than 15 years or less than 50 kg if age unknown
* Ongoing pre-hospital cardiopulmonary resuscitation (CPR)
* Administration of more than 2L crystalloid or any colloid or blood products
* Severe hypothermia (T less than 28C)
* Drowning or asphyxia due to hanging
* Burns TBSA more than 20%
* Isolated penetrating injury to the head
* Inability to obtain pre-hospital intravenous access
* Time of call received at dispatch to study intervention more than four hours
* Known prisoners

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1331 (Actual)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron L Weisfeldt, MD, Study Chair — Resuscitation Outcomes Consortium
Locations (12):
- United States (10):
  - Alabama Resuscitation Center, University of Alabama, Birmingham, Alabama
  - Orange County/UC Irvine, Orange, California
  - UCSD-San Diego Resuscitation Research Center, San Diego, California
  - Iowa Resuscitation Network, University of Iowa Carver College of Medicine, Iowa City, Iowa
  - Portland Resuscitation Outcomes Consortium, Oregon Health & Sciences University, Portland, Oregon
  - The Pittsburgh Resuscitation Network, University of Pittsburgh, Pittsburgh, Pennsylvania
  - The Regional Medical Center at Memphis, Memphis, Tennessee
  - Dallas Center for Resuscitation Research, University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle-King County Center for Resuscitation Research, University of Washington, Seattle, Washington
  - Milwaukee Resuscitation Network, Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - University of Ottawa/University of British Columbia Collaborative RCC, Ottawa Health Research Institute, Ottawa, Ontario
  - Toronto Regional Resuscitation Research Out-of-Hospital Network, University of Toronto, Toronto, Ontario

REFERENCES:
- [Result] Bulger EM, May S, Brasel KJ, Schreiber M, Kerby JD, Tisherman SA, Newgard C, Slutsky A, Coimbra R, Emerson S, Minei JP, Bardarson B, Kudenchuk P, Baker A, Christenson J, Idris A, Davis D, Fabian TC, Aufderheide TP, Callaway C, Williams C, Banek J, Vaillancourt C, van Heest R, Sopko G, Hata JS, Hoyt DB; ROC Investigators. Out-of-hospital hypertonic resuscitation following severe traumatic brain injury: a randomized controlled trial. JAMA. 2010 Oct 6;304(13):1455-64. doi: 10.1001/jama.2010.1405. PMID 20924011
- [Derived] Tisherman SA, Schmicker RH, Brasel KJ, Bulger EM, Kerby JD, Minei JP, Powell JL, Reiff DA, Rizoli SB, Schreiber MA. Detailed description of all deaths in both the shock and traumatic brain injury hypertonic saline trials of the Resuscitation Outcomes Consortium. Ann Surg. 2015 Mar;261(3):586-90. doi: 10.1097/SLA.0000000000000837. PMID 25072443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled by Emergency Medicine Services (EMS) personnel in the prehospital setting based on pre-defined inclusion/exclusion criteria. The first subject was enrolled in May 2006. The last subject was enrolled in May 2009.
Pre-assignment Details: 1331 subjects were randomized. 1282 were included in primary imputation analysis. 49 were randomized with study fluid package opened but no study fluid was given. Reasons given were: Did not meet inclusion criteria; Met an exclusion criterion; No intravenous access; Fluid bag sterility broken; EMS responder unsure of inclusion/exclusion criteria.
Groups:
- 7.5% Hypertonic Saline/6% Dextran (HSD): 250 ml intravenous bolus administration of 7.5% saline/6% dextran 70 as the initial resuscitation fluid given to injured patients with suspected severe traumatic brain injury in the out-of-hospital setting.
- 7.5% Hypertonic Saline (HS): 250 ml intravenous bolus administration of 7.5% hypertonic saline as the initial resuscitation fluid given to injured patients with suspected severe traumatic brain injury in the out-of-hospital setting.
- 0.9% Normal Saline (NS): 250 ml intravenous bolus administration of 0.9% saline as the initial resuscitation fluid given to injured patients with suspected severe traumatic brain injury in the out-of-hospital setting.
Period: Overall Study
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Started | 373 | 355 | 603
Completed | 359 | 341 | 582
Not Completed | 14 | 14 | 21
Not completed — Subject was not given study fluid. | 14 | 14 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS) | Total
Number analyzed (Participants) | 373 | 355 | 603 | 1331
Age Categorical [Number; unit: participants] — The HSD group included 3 subjects with no age data available. The HS group included 2 subjects with no age data available. The NS group included 2 subjects with no age data available.
  participants
    <=18 years | 33 | 19 | 43 | 95
    Between 18 and 65 years | 296 | 305 | 484 | 1085
    >=65 years | 41 | 29 | 74 | 144
Age Continuous [Mean (Standard Deviation); unit: years] — The HSD group included 3 subjects with no age data available. The HS group included 2 subjects with no age data available. The NS group included 2 subjects with no age data available.
  years | 38.5 (18.6) | 38.6 (17.3) | 39.5 (19.2) | 39.0 (18.4)
Gender [Number; unit: participants] — The HSD group included 3 subjects with no gender data available. The HS group included 1 subject with no gender data available. The NS group included 2 subjects with no gender data available.
  participants
    Female | 86 | 68 | 163 | 317
    Male | 284 | 286 | 438 | 1008
Region of Enrollment [Number; unit: participants]
  United States | 291 | 259 | 441 | 991
  Canada | 82 | 96 | 162 | 340

OUTCOME MEASURES:

1. Primary Outcome: Glasgow Outcome Scale-Extended (GOSE)≤4 at 6 Months: Completer Analysis
Description: Glasgow outcome score extended (GOSE) contains eight categories: 1. Dead, 2. Vegetative State (VS), 3. Lower Severe Disability (Lower SD), 4. Upper Severe Disability (Upper SD), 5. Lower Moderate Disability (Lower MD), 6. Upper Moderate Disability (Upper MD), 7. Lower Good Recovery (Lower GR) and 8. Upper Good Recovery (Upper GR). A measured neurological outcome of GOSE≤4 is a poor outcome of severe disability, vegetative state, or death. Completer analysis includes only those patients with GOSE completed at 6 months after injury.
Time Frame: 6 months after injury
Population: The primary analysis was designed as modified intent-to-treat, with all patients who had fluid connected to intravenous (IV) tubing included regardless of how much fluid was administered. Per the a priori trial design, patients for whom the fluid bag was opened but not connected to the IV were not considered enrolled in the trial.
Measure: Number; unit: Participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 302 | 293 | 492
Participants | 181 | 171 | 276
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent prevalence of poor outcome between the three groups; Test type: Superiority or Other; p = 0.55, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups

2. Secondary Outcome: Subgroup of Participants With Head Abbreviated Injury Scores (AIS) Greater Than or Equal to 4 (Head AIS≥4) Assessed to Have Glasgow Outcome Scale-Extended (GOSE)≤4 at 6 Months: Imputed Analysis
Description: The Abbreviated Injury Scale (AIS) ranks injuries on a scale of 1 to 6, with 1 being minor, 2 moderate, 3 serious, 4 severe, 5 critical and 6 an unsurvivable injury. A priori secondary analyses included the subgroup of participants in each intervention group with a head AIS≥4, which is a diagnostic indicator of severe to lethal head injury. Of this subset of participants with AIS≥4, a second subset of participants with a GOSE≤4 at the 6 month follow up was analyzed. GOSE≤4 represents Upper Severe Disability or worse outcomes. 15% of subjects required imputation analysis for 6-month GOSE.
Time Frame: 6 months after injury
Population: To adjust for 15% of subjects with absent 6-month GOSE data, an analysis using 20 hot deck imputations for the 6-month GOSE was done using data from patients who were discharged alive based on 1-month post discharge GOSE data or discharge GOSE (if 1-month post discharge data were not available), length of hospital stay, and treatment group.
Measure: Number; unit: Participants (with imputed values)
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 208 | 193 | 331
Participants (with imputed values) | 146.1 | 128.0 | 219.0
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent prevalence of poor outcome between the three treatment groups among patients with head AIS≥4; Test type: Superiority or Other; p = 0.59, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups; Adjusted for multiple imputations

3. Primary Outcome: Glasgow Outcome Scale-Extended (GOSE)≤4 at 6 Months: Imputed Analysis
Description: Glasgow outcome score extended (GOSE) contains 8 categories: 1. Dead, 2. Vegetative State, 3. Lower Severe Disability, 4. Upper Severe Disability, 5. Lower Moderate Disability, 6. Upper Moderate Disability, 7. Lower Good Recovery and 8. Upper Good Recovery. To adjust for 15% of subjects with absent 6-month GOSE data, an analysis using 20 hot deck imputations for the 6-month GOSE was done using data from patients who were discharged alive based on 1-month post discharge GOSE data or discharge GOSE (if 1-month post discharge data were not available), length of hospital stay, and treatment group.
Time Frame: 6 months after injury
Population: as for outcome 2
Measure: Number; unit: Participants (with imputed values)
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 359 | 341 | 582
Participants (with imputed values) | 192.9 | 185.4 | 299.8
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent prevalence of poor outcome between the three groups; Test type: Superiority or Other; p = 0.67, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups; Adjusted for multiple imputations

4. Secondary Outcome: Subgroup of Participants With Head Abbreviated Injury Scores (AIS) Greater Than or Equal to 2 (Head AIS≥2) Assessed to Have Glasgow Outcome Scale-Extended (GOSE)≤4 at 6 Months: Imputed Analysis
Description: The Abbreviated Injury Scale (AIS) ranks injuries on a scale of 1 to 6, with 1 being minor, 2 moderate, 3 serious, 4 severe, 5 critical and 6 an unsurvivable injury. A priori secondary analyses included the subgroup of participants in each intervention group with a head AIS≥2, which is a diagnostic indicator of moderate to lethal head injury. Of this subset of participants with AIS≥2, a second subset of participants with a GOSE≤4 at the 6 month follow up was analyzed. GOSE≤4 represents Upper Severe Disability or worse outcomes. 15% of subjects required imputation analysis for 6-month GOSE.
Time Frame: 6 months after injury
Population: as for outcome 2
Measure: Number; unit: Participants (with imputed values)
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 281 | 268 | 458
Participants (with imputed values) | 166.7 | 150.6 | 253.2
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent prevalence of poor outcome between the three treatment groups among patients with head AIS≥2; Test type: Superiority or Other; p = 0.57, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups; Adjusted for multiple imputations

5. Secondary Outcome: Disability Rating Score (DRS) Categories of Disability
Description: The DRS is an additional measure of neurological outcome that categorizes the patient's level of disability on a scale of 0 to 29, with 0 indicating no disability to 29 indicating extreme vegetative state. To adjust for 15% of subjects with absent 6-month DRS data, an analysis using 20 hot deck imputations for the 6-month DRS was done using data from patients who were discharged alive based on 1-month post discharge DRS data or discharge DRS (if 1-month post discharge data were not available), length of hospital stay, and treatment group.
Time Frame: 6 months after injury
Population: To adjust for 15% of subjects with absent 6-month DRS data, an analysis using 20 hot deck imputations for the 6-month DRS was done using data from patients who were discharged alive based on 1-month post discharge DRS data or discharge DRS (if 1-month post discharge data were not available), length of hospital stay, and treatment group.
Measure: Number; unit: Participants (with imputed values)
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 359 | 341 | 582
Participants (with imputed values)
  0-1 (none/mild disability) | 124.8 | 128.0 | 232.0
  2-6 (Partial/Moderate Disability) | 98.3 | 89.4 | 143.2
  7-21 (moderately severe/severe/extremely severe) | 33.0 | 26.6 | 43.3
  22-30 (vegetative/extreme vegetative/dead) | 102.9 | 97.0 | 163.4
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients at any level of disability between the three groups; Test type: Superiority or Other; p = .84, test for proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups; Adjusted for multiple imputations

6. Secondary Outcome: 28 Day Survival
Description: The patient who is admitted to the hospital after injury and is alive on the 28th day after injury. For 28-day survival, patients with missing 28-day vital status who were known to be discharged alive prior to 28 days were assumed to be alive at day 28.
Time Frame: 28 days after injury
Population: An analysis of this secondary outcome was done for all participants assigned to each of the three groups who did not refuse or were lost to follow-up prior to discharge.
Measure: Number; unit: Participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 357 | 340 | 575
Participants | 268 | 260 | 432
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients who were alive on the 28th day after injury between the three groups; Test type: Superiority or Other; p = 0.88, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups; The numbers differ from the JAMA manuscript because of typos and version control issues that were discovered after publication

7. Secondary Outcome: Survival at Hospital Discharge up to 6 Months From Date of Injury
Description: The patient who is admitted to the hospital alive after injury and is alive when discharged from the hospital up to 6 months from the date of injury.
Time Frame: Date of hospital discharge up to 6 months from date of injury
Population: An analysis of this secondary outcome was done for all participants assigned to each of the three groups who had relevant data.
Measure: Number; unit: Participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 354 | 337 | 575
Participants | 263 | 255 | 427
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients who were alive on the day discharged from the hospital after injury between the three groups; Test type: Superiority or Other; p = 0.88, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups; [statistical method as in outcome 6, analysis 1]

8. Secondary Outcome: Acute Respiratory Distress Syndrome (ARDS)-Free Survival to Day 28
Description: The patient is alive and free of ARDS from the date of injury through to the 28th day following injury. The diagnosis of ARDS is based on standard criteria: a) hypoxia with a ratio of arterial oxygen pressure to percent oxygen delivered of less than 200; b) bilateral infiltrates on chest X-ray; and c) clinical evidence of increased left atrial pressure or pulmonary artery wedge pressure of greater than 18 mmHg.
Time Frame: From day of injury to 28 days after injury
Population: Number of participants analyzed in each group is the actual number analyzed, which does not include participants with one of the following: 1. prehospital death; 2. transfer to another hospital without IRB approval; or 3. patient, family member, or legally authorized representative refused consent and was withdrawn from the study.
Measure: Number; unit: Participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 356 | 337 | 572
Participants | 247 | 239 | 401
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients who were alive and free of ARDS from the day of injury to the 28th day after injury between the three groups; Test type: Superiority or Other; p = 0.91, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups; [statistical method as in outcome 6, analysis 1]

9. Secondary Outcome: Worst Multiple Organ Dysfunction Score (MODS) Through Day 28
Description: Multiple Organ Dysfunction Score is described as: Six organ systems were chosen: 1) respiratory; 2) renal; 3) hepatic; 4) cardiovascular; 5) hematologic; and 6) neurologica. A score of 0-4 was allotted for each organ according to function (0 being normal function through 4 for most severe dysfunction) with a maximum score of 24. The worst score based on available data (missing values were assumed normal) was taken for calculation of the aggregate score. Deaths are assigned the worst score (24).
Time Frame: From day of injury to 28 days after injury
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 348 | 329 | 558
Scores on a scale | 9 (9.3) | 8.6 (9.3) | 8.6 (9.5)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in average Worst Multiple Organ Dysfunction Scores (MODS) through day 28 between the three groups; Test type: Superiority or Other; p = 0.81, ANOVA — The p-value was not adjusted for multiple comparisons. Test compares averages across all three treatment groups; [statistical method as in outcome 6, analysis 1]

10. Secondary Outcome: Ventilator-free Days Through Day 28
Description: The number of days beginning with the day of 911 call counted as "Day 0" through day 28 that the patient did not require mechanical ventilation. Deaths are assigned the worst score (0).
Time Frame: From day of injury to 28 days after injury
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 355 | 337 | 572
Days | 17.0 (11.6) | 17.6 (11.5) | 17.4 (11.7)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the average number of Ventilator-free days through day 28 between the three groups; Test type: Superiority or Other; p = 0.77, ANOVA — The p-value was not adjusted for multiple comparisons. Test compares averages across all three treatment groups; [statistical method as in outcome 6, analysis 1]

11. Secondary Outcome: Days Alive Out of the Intensive Care Unit (ICU) Through Day 28
Description: The number of days the patient is alive and not being cared for in the intensive care unit
Time Frame: From day of injury to 28 days after injury
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 355 | 337 | 572
Days | 15.2 (11.5) | 15.8 (11.4) | 15.6 (11.7)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the average number of days alive out of the ICU through day 28 between the three groups; Test type: Superiority or Other; p = 0.76, ANOVA — The p-value was not adjusted for multiple comparisons. Test compares averages across all three treatment groups; [statistical method as in outcome 6, analysis 1]

12. Secondary Outcome: Days Alive Out of the Hospital Through Day 28
Description: The number of days the patient is alive and no longer an inpatient in the hospital through day 28
Time Frame: From day of injury to 28 days after injury
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 354 | 337 | 575
Days | 9.8 (10.9) | 10 (11.0) | 10.7 (11.2)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the average number of days alive out of the hospital through day 28 between the three groups; Test type: Superiority or Other; p = 0.43, ANOVA — The p-value was not adjusted for multiple comparisons. Test compares averages across all three treatment groups; [statistical method as in outcome 6, analysis 1]

13. Secondary Outcome: Presence of Nosocomial Infections
Description: Includes one or more nosocomial infections diagnosed during the hospital stay but not present on admission to the hospital from the following list: pneumonia, bloodstream infection, urinary tract infection, and/or wound infection
Time Frame: From day of injury to 28 days after injury
Population: An analysis of this secondary outcome was done for all participants assigned to each of the three groups who had relevant data. Percentages were based on population at risk.
  Row 1 nosocomial infections; Row 2 pneumonia; Row 3 bloodstream infections; Row 4 urinary tract infections; and Row 5 wound infections
Measure: Number; unit: Diagnoses
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 320 | 313 | 530
Diagnoses
  Nosocomial Infections ≥ 1 | 102 | 101 | 136
  Pneumonia | 72 | 71 | 100
  Bloodstream Infection | 23 | 21 | 19
  Urinary Tract Infection | 30 | 32 | 32
  Wound Infection | 8 | 8 | 16
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients with any nosocomial infections through hospital stay between the three groups; Test type: Superiority or Other; p = 0.06, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups
Statistical Analysis 2: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients with pneumonia through hospital stay between the three groups; Test type: Superiority or Other; p = 0.3, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups
Statistical Analysis 3: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients with bloodstream infections through hospital stay between the three groups; Test type: Superiority or Other; p = 0.04, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups
Statistical Analysis 4: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients with urinary tract infections through hospital stay between the three groups; Test type: Superiority or Other; p = 0.06, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups
Statistical Analysis 5: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients with wound infections through hospital stay between the three groups; Test type: Superiority or Other; p = 0.88, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups

14. Secondary Outcome: Total Fluids in First 24 Hours
Description: The average (mean) total amount of intravenous (IV) fluids given in the pre-hospital setting and the hospital setting in the first 24 hours following the time of the 911 call
Time Frame: First 24 hours from the time dispatch received 911 call
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 357 | 341 | 581
Liters | 6.7 (5.5) | 6.7 (5.5) | 6.9 (5.7)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the average amount of total fluids given within the first 24 hours between the three groups; Test type: Superiority or Other; p = 0.68, ANOVA — The p-value was not adjusted for multiple comparisons. Test compares averages across all three treatment groups

15. Secondary Outcome: Packed Red Blood Cells (PRBC) First 24 Hours
Description: The average (mean) number of units of packed red blood cells (PRBC) transfused in the first 24 hours following the time of the 911 call in each group.
Time Frame: First 24 hours from the time dispatch received 911 call
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Unit of PRBC
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 356 | 341 | 580
Unit of PRBC | 1.4 (3.6) | 1.2 (3.4) | 1.5 (4.3)
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the average number of PRBC units given within the first 24 hours between the three groups; Test type: Superiority or Other; p = 0.43, ANOVA — The p-value was not adjusted for multiple comparisons. Test compares averages across all three treatment groups

16. Secondary Outcome: Discharge Disposition
Description: Disposition of patient at the time of discharge from the acute care hospital
Time Frame: Duration of hospital stay
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Number analyzed (Participants) | 352 | 336 | 574
Participants
  Death | 89 | 81 | 147
  Home | 138 | 134 | 253
  Inpatient Rehabilitation | 84 | 90 | 122
  Skilled Nursing Facility | 37 | 28 | 40
  Nursing Home or Inpatient Psychiatric Facility | 4 | 3 | 12
Statistical Analysis 1: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients who died during hospitalization between the three groups; Test type: Superiority or Other; p = 0.88, test for proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups
Statistical Analysis 2: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients who were discharged alive from the hospital to home between the three groups; Test type: Superiority or Other; p = 0.26, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups
Statistical Analysis 3: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients who were discharged alive from the hospital to inpatient rehabilitation facilities between the three groups; Test type: Superiority or Other; p = 0.16, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups
Statistical Analysis 4: Comparison: 7.5% Hypertonic Saline/6% Dextran (HSD) vs 7.5% Hypertonic Saline (HS) vs 0.9% Normal Saline (NS); The null hypothesis is that there are no differences in the percent of patients who were discharged alive from the hospital to skilled nursing facilities between the three groups; Test type: Superiority or Other; p = 0.17, test for differences in proportions — The p-value was not adjusted for multiple comparisons. Test compares proportions across all three treatment groups

ADVERSE EVENTS:
Time Frame: The time frame was from May 2006 through May 2009, which was 3 years
Description: Serial blood sodium levels were drawn to monitor the effects of the hypertonic saline solutions; Serial head CT's (computed tomography) were done to monitor for increased intracranial hemorrhage; and incidents of seizures in the first 24 hours.
Arm/Group | 7.5% Hypertonic Saline/6% Dextran (HSD) | 7.5% Hypertonic Saline (HS) | 0.9% Normal Saline (NS)
Serious Adverse Events (participants affected / at risk) | 69/359 | 72/341 | 141/582
Other Adverse Events (participants affected / at risk) | 0/359 | 0/341 | 0/582
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 7.5% Hypertonic Saline/6% Dextran (HSD) (N=359) | 7.5% Hypertonic Saline (HS) (N=341) | 0.9% Normal Saline (NS) (N=582)
Hypernatremia (sodium>160 mEq/L) requiring intervention (Blood and lymphatic system disorders) | 10/349 (10) | 14/334 (14) | 13/573 (13) — Hypernatremia (sodium>160 mEq/L) requiring intervention to decrease serum sodium level to prevent additional complications.
Increased intracranial hemorrhage on serial head CT (Nervous system disorders) | 57/349 (57) | 60/325 (60) | 122/560 (122) — Increased intracranial hemorrhage on serial head CT was observed.
Seizures in the first 24 hours (Nervous system disorders) | 4 (4) | 3 (3) | 12 (12) — Incidents of seizures observed in the first 24 hours

LIMITATIONS AND CAVEATS:
The trial was stopped early for futility at a planned data and safety monitoring board review. The futility boundary was crossed for each of the 2 group comparisons (hypertonic saline/dextran vs normal saline and hypertonic saline vs normal saline).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No